CLINICAL TRIAL: NCT00909766
Title: Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple-Dose and Parallel Arm Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-830216 (Prodrug of BMS-819881) in Obese Subjects
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics Study to Evaluate BMS-830216 in Obese Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB123-002
Record Dates: First submitted 2009-05-22; First posted 2009-05-28 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Panel A (Active Comparator)
  Interventions: Drug: BMS-830216; Drug: Placebo
- Panel B (Active Comparator)
  Interventions: Drug: BMS-830216; Drug: Placebo
- Panel C (Active Comparator)
  Interventions: Drug: BMS-830216; Drug: Placebo
- Panel D (Active Comparator)
  Interventions: Drug: BMS-830216; Drug: Placebo
- Panel E (Active Comparator)
  Interventions: Drug: BMS-830216; Drug: Placebo
- Panel F (Active Comparator): Low Dose
  Interventions: Drug: BMS-830216
- Panel G (Active Comparator): High Dose
  Interventions: Drug: BMS-830216
- Panel H (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-830216 — Capsules, Oral, 30 mg, once daily, 28 days
  Arms: Panel A
Drug: BMS-830216 — Capsules, Oral, 100 mg, once daily, 28 days
  Arms: Panel B
Drug: BMS-830216 — Capsules, oral, 300 mg, once daily, 28 days
  Arms: Panel C
Drug: BMS-830216 — Capsules, oral, 600 mg, once daily 28 days
  Arms: Panel D
Drug: BMS-830216 — Capsules, oral, 1200 mg, once daily, 28 days
  Arms: Panel E
Drug: BMS-830216 — Capsules, Oral, to be determined, once daily, 28 days
  Arms: Panel F; Panel G
Drug: Placebo — Capsules, Oral, 0 mg, once daily, 28 days
  Arms: Panel A; Panel B; Panel C; Panel D; Panel E; Panel H

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and effect on body weight and other obesity-related factors of different doses of BMS-830216, compared to placebo. The study will also determine the amount of BMS-830216 in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body Mass Index (BMI) of 30 to 40 kg/m², inclusive
* Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) and men, ages 18 to 55, inclusive

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population
* Female of childbearing potential
* Sexually active fertile male not using effective birth control method (for example, condom) if your partners are females of childbearing potential
* Abnormal blood work results (for example, triglyceride ≥ 400 mg/dL, glucose ≥126 mg/dL and total cholesterol ≥ 300 mg/dL)
* High blood pressure (≥160/95 mm Hg)
* Major surgical procedure within 4 weeks prior to randomization
* Chronic infections (e.g., HIV [human immunodeficiency virus] or Hepatitis C)
* Clinically significant history or presence of any of the following conditions: heart, liver, or kidney disease, neurologic or psychiatric disease, or a previous surgery for weight loss
* History of gastrointestinal disease within the past 3 months
* History of Type I or Type II diabetes in the past 12 months
* A lifetime history of a suicide attempt or history of any suicidal behavior in the past month
* Any clinically significant medical condition that could potentially affect your participation in the study and/or personal well-being, as judged by the investigator
* Used grapefruit or grapefruit juice within 1 week prior to randomization
* Donated blood or blood products to a blood bank, blood transfusion or participated in a clinical study (except a screening visit) requiring withdrawal of blood within 4 weeks prior to randomization
* Unable to tolerate oral and/or intravenous (IV) medications
* Unable to tolerate the puncturing of veins for drawing of blood
* Prior exposure to BMS-830216
* History of prior weight loss (for example, gastric bypass or gastric banding) or gastrointestinal surgery that could impact the absorption of study drug
* History of a Major Depressive Disorder within the past 2 years
* Known allergy or hypersensitivity to any component of the study medication
* History of any significant drug allergies (such as anaphylaxis or hepatotoxicity)
* Used any oral, injectable or implantable hormonal contraceptive agents (for example, birth control pills, Depo-Provera, or NuvaRing) within 3 months prior to randomization
* Used any prescription drugs or over the counter products to control acid (for example, Prevacid, Mylanta or Rolaids) within 4 weeks prior to randomization
* Used any prescription drugs, over the counter medications and herbal preparations within 1 week prior to randomization
* Taken St. John's Wort within 1 week prior to randomization
* Taken any investigational drug or placebo (inactive drug) within 4 weeks prior to randomization

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety: safety assessments will be based on adverse event reports and the results of vital sign measurements, electrocardiograms, physical examinations and clinical laboratory tests | Within 2 weeks after study drug administration

SECONDARY OUTCOMES:
Pharmacokinetics: to assess the multiple-dose PK of BMS-830216 | Within 2 weeks of study drug administration
Pharmacodynamics: to assess the pharmacodynamic effect of BMS-830216 on body weight and BMI over 4 weeks of therapy | Within 2 weeks of study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx